CLINICAL TRIAL: NCT02355977
Title: The Response of Periodontal Pathogens to the Respective or Combined Treatment of Scaling and Root Planning and Locally Delivered Minocycline in Patients With Chronic Periodontitis- a Short-term Randomized Clinical Trial
Brief Title: The Response of Pathogens to the Respective or Combined Treatment of SRP and Local Minocycline in Chronic Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Shuli Deng, Dr., Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-25
Record Dates: First submitted 2015-01-31; First posted 2015-02-04 (Estimated); Results first posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Minocycline; Surface and root planning; Pocket depth; Sulcus bleeding index; Prevotella intermedia
MeSH Terms: conditions — Chronic Periodontitis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- surface and root planning (Active Comparator): surface and root planning is performed in a single-visit, one-stage, full mouth pattern using periodontal ultrasonic scaler (Satelec, Mérignac, France)
  Interventions: Procedure: surface and root planning
- locally delivered minocycline (Active Comparator): Locally delivered minocycline is administered directly into the periodontal pocket up to the gingival margin of the selected teeth
  Interventions: Drug: minocycline; Procedure: surface and root planning
- surface and root planning+minocycline (Experimental): surface and root planning+locally delivered minocycline is the combined administration of both surface and root planning and locally delivered minocycline.
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — Periocline dental ointment
  Other Names: Periocline dental ointment
  Arms: locally delivered minocycline; surface and root planning+minocycline
Procedure: surface and root planning — surface and root planning
  Arms: locally delivered minocycline; surface and root planning

SUMMARY:
To evaluate the respective or combinatory efficacy of locally delivered 2% Minocycline (MO) and surface and root planning (SRP) by assessing both clinical parameters and the loads of four main periodontal pathogens in treating chronic periodontitis.

DETAILED DESCRIPTION:
In this randomized clinical trial, the investigators will evaluate the respective or combinatory efficacy of minocycline and scaling and root planning in the aspects of both clinical parameters [Pocket depth (PD) and sulcus bleeding index (SBI)] and the loads of four main periodontal pathogens [Aggregatibacter actinomycetemcomitans (Aa), Fusobacterium nucleatum (Fn), Porphyromonas gingivalis (Pg) and Prevotella intermedia (Pi)]. Real-time quantitative PCR (qRT-PCR) will be used as a powerful tool with high sensitivity and specificity to quantitatively assess target periodontal bacteria in a period of 7 days. The investigators will also try to correlate the reduction of either total or respective bacteria with the improvements of clinical parameters, with an aim to uncovering the potential microbiological mechanism accounting for the efficacy of a therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with moderate or severe chronic periodontal disease, and exhibited bleeding on probing and attachment loss, with radiographic alveolar bone loss in four or more teeth

Exclusion Criteria:

* pregnant, had used antibiotics within the last 3 months, had periodontal therapy in the past 6 months or had systemic diseases such as heart disease or hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuli Deng, Master, Principal Investigator — Affiliated Hospital of Stomatology, Medical College, Zhejiang University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline
Started | 21 | 26 | 23
Completed | 21 | 26 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline | Total
Number analyzed (Participants) | 21 | 26 | 23 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 22 | 64
  >=65 years | 1 | 4 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15) | 50 (13) | 49 (11) | 49 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 12 | 34
  Male | 8 | 17 | 11 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 26 | 23 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 21 | 26 | 23 | 70

OUTCOME MEASURES:

1. Primary Outcome: Pocket Depth
Description: PD is measured using a standard CPI（community periodontal index） probe (Shanghai Medical Instruments, Shanghai, China) and assessed to the nearest millimeter.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline
Number analyzed (Participants) | 21 | 26 | 23
mm | 4.34 (0.57) | 4.81 (0.99) | 4.5 (0.53)

2. Secondary Outcome: Bleeding on Probing
Description: BOP is evaluated for the treated tooth using the sulcus bleeding index (SBI) by Muhlemann with a range of 0 (no bleeding) to 5 (profuse bleeding)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline
Number analyzed (Participants) | 21 | 26 | 23
units on a scale | 1.42 (0.55) | 1.23 (0.70) | 1.42 (0.55)

3. Secondary Outcome: Bacterial Load
Description: Real-time quantitative PCR (qRT-PCR) was used as a powerful tool with high sensitivity and specificity to quantitatively assess target periodontal bacteria.
Time Frame: 7 days
Population: The analyzed units of the gene load of bacteria are log10.
Measure: Mean (Standard Deviation); unit: log10 (copies/ml)
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline
Number analyzed (Participants) | 21 | 26 | 23
log10 (copies/ml)
  Aggregatibacter actinomycetemcomitans (Aa) | 5.55 (0.59) | 4.32 (1.67) | 4.77 (0.86)
  Fusobacterium nucleatum (Fn) | 6.77 (0.39) | 6.37 (0.43) | 6.72 (0.42)
  Porphyromonas gingivalis (Pg) | 7.11 (1.77) | 6.72 (1.73) | 7.13 (1.78)
  Prevotella intermedia (Pi) | 4.98 (0.72) | 4.58 (1.16) | 4.77 (0.92)

ADVERSE EVENTS:
Arm/Group | Surface and Root Planning | Locally Delivered Minocycline | Surface and Root Planning+Minocycline
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 0/26 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes